CLINICAL TRIAL: NCT03479398
Title: Leveraging Routine Clinical Materials and Mobile Technology to Assess CBT Quality
Brief Title: Innovative Methods to Assess Psychotherapy Practices (imAPP)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Shannon Wiltsey Stirman, Psychologist/Implementation Scientist, Palo Alto Veterans Institute for Research
Other Study IDs: WIS0003AGG; R01MH112628 (NIH)
Record Dates: First submitted 2018-03-08; First posted 2018-03-27 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Mobile Application-Based CBT Worksheet Collection; Paper-Based Worksheet Collection
Keywords: Fidelity; Cognitive Behavioral Therapy; Mobile Application; Routine Practice
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- App Condition: Although we will be mostly observing routine practice, we will randomize patients into either an App condition or paper condition. The App condition refers to patients completing routine Cognitive Behavioral Therapy (CBT) worksheets on a mobile application during session. Everything else that occurs in treatment sessions will be consistent with routine care practices.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Paper Condition: Although we will be mostly observing routine practice, we do randomize patients into either an App condition or paper condition. The paper condition refers to patients completing routine CBT worksheets on paper (the current standard) during session.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy (CBT) is an evidence-based psychotherapy that treats a variety of disorders. In this study, clinicians will be enrolled who use types of CBT for anxiety disorders, depression and PTSD in their routine clinical practice. CBT is usually a 12-16 session treatment that focuses on intervening on disorders cognitively and behaviorally through the use of worksheets during session and outside of session.
  Other Names: Cognitive Processing Therapy

SUMMARY:
This project compares two methods of assessing the quality of cognitive behavioral therapy (CBT) that do not involve directly observing sessions: 1) adherence checklists embedded in clinical notes, and 2) rating the quality of worksheets that are completed with therapist guidance during sessions. It also examines whether ratings of worksheets completed on a mobile app are reliable and valid quality measures. This information can inform strategies to monitor and enhance CBT quality, which can ultimately improve the quality of care and clinical outcomes.

DETAILED DESCRIPTION:
Cognitive Behavioral Therapy (CBT) has been demonstrated to be effective for numerous presenting problems, including depression, anxiety, and post-traumatic stress disorder (PTSD). Several large mental health systems have invested heavily in programs to train their clinicians in CBTs, but relatively little attention has been devoted to the monitoring or promotion of CBT quality after training is complete. Identifying strategies to do so can facilitate research and training, and is critical to ensuring consumer access to high quality, evidence-based treatments. The lack of a scalable, effective, and efficient method of monitoring quality is a key barrier to efforts to promote high-quality implementation. Self-report fidelity assessments increase clinician and consumer burden and may not accurately reflect clinician skill or the intensity with which CBT interventions are delivered. Observation and expert ratings are time and resource intensive and unlikely to be feasible or affordable in large systems. To maximize the likelihood of broad implementation once effective strategies to monitor quality are established, it is essential that these strategies are feasible and acceptable in routine care contexts, leveraging information collected during routine care. To date, few monitoring strategies that do not involve observation, client/caregiver reports, or clinician self-reports have been tested. To address this critical implementation challenge, we propose to refine and evaluate a method of monitoring quality that is based on an evaluation of CBT worksheets that are completed in session. Because the worksheets were developed to implement core cognitive and behavioral elements and are embedded in CBTs across diagnostic categories, they may be used to elucidate the clinician's ability to guide the client through CBT interventions in session. Preliminary research with this measure demonstrated high correlations between the measure and observer ratings of clinician competence, associations with subsequent symptom change, and high agreement between raters with differing levels of familiarity with CBT. Completion of the ratings based on worksheets requires only a small fraction of time required for session observation and ratings. This project will compare this novel strategy to observer ratings and adherence checklists that are embedded in clinical notes. Furthermore, it will compare the accuracy of worksheet data collected by mobile app to paper-form worksheets, and assess the feasibility and acceptability of these strategies. Because the core elements of CBT and its worksheets are common across many CBTs, this research has broad implications for monitoring fidelity to CBTs in a variety of mental health and healthcare systems and settings. This research will be conducted by a team of investigators with expertise in CBT, training, implementation, psychotherapy process and outcome research, psychometrics, longitudinal data analysis, mobile technologies and healthcare economics, with input from community partners and end-users. The resulting products have the potential to significantly improve efforts to monitor and ensure ongoing high quality implementation of CBT in routine care settings.

ELIGIBILITY:
Inclusion Criteria:

A. Clinician eligibility:

* Private practice or employment at an agency at which the administration agrees to allow the recruitment and participation of their providers in research related activities
* English Speaking
* No anticipated plans to leave their current agency for at least 18 months
* Willingness to allow their CBT sessions, worksheets, surveys, and interview data, and clinical notes to be used for research purposes
* Carry a caseload that typically includes patients who experience depression, anxiety, or PTSD, with whom they regularly conduct individual therapy sessions and/or capacity to increase the proportion of such patients (e.g., clinic sees a substantial number of individuals with PTSD or depression)
* Must be trained (worksheet or web-based training and consultation) or in training for Cognitive Processing Therapy (CPT) for PTSD or CBT for depression or anxiety that uses worksheets Does not include CBT-i Can include aspects (i.e., worksheets) of CBT for substance use as long as depression or anxiety is primary diagnoses
* Must anticipate at least 3 eligible patients
* Must be willing to record sessions and provide worksheets and symptom measures to the study
* Must have computer and internet access
* Must be willing to use a mobile app on a tablet or mobile device

B. Patient eligibility:

* Must be 18 yrs. of age or older
* Experience one or more of the following (both a diagnosis and cut off score):

Clinician diagnosis of primary PTSD (PTSD-Checklist-5 score of 33 or more) Depressive disorder (e.g., major depressive disorder, dysthymia; PHQ of 10 or above) Or an Anxiety Disorder (Beck Anxiety Disorder score of 22 or above)

* Note that if a patient has a score close to the cut-off score, it's up to the therapist digression

  * Must be willing to allow the team to collect session recordings, measures, notes and worksheets
  * Must be able to read and write at a sixth-grade level or above
  * Able to participate in sessions conducted in English, or Spanish (if working with bilingual clinicians in community or private practice)
  * Must be willing to engage in CBT/CPT
  * Therapist considers the treatment with the individual patient to be "mostly" CBT or CPT

Cannot have*:

- Imminent risk of suicide or homicide (requiring hospitalization) that require immediate treatment In need of detoxification (can be enrolled when substance abuse treatment is not the primary treatment target) Active psychosis or manic episode unless well controlled by medication and not the primary focus of treatment Cognitive impairments that preclude any participation in therapy

C. Administrator eligibility:

* Must have a support or managerial/supervisory position at the clinic(s) from which A and B are being recruited from
* Must also be willing to complete a packet of study measures/partake in an interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Therapists who provide Cognitive Behavioral Therapy, and their patients who receive CBT for depression, anxiety, or PTSD. Therapists and patients will be recruited from community-based, public mental health (e.g., Boston and Palo Alto VA) and private practice treatment settings.
Sampling Method: Probability Sample
Enrollment: 439 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-9) | Baseline (pre-treatment), Every session (weekly) if primary /target problem up to 16 weeks
  9-item self-report measure of depression symptoms with good internal reliability (α = .89) and test-retest reliability (r = .84).
Change in Posttraumatic Stress Disorder Checklist (PCL-5) | Baseline (pre-treatment), Every session (weekly) if primary /target problem up to 16 weeks
  A 20-item self-report measure that assesses the 20 Diagnostic and Statistical Manual (DSM-5) symptoms of PTSD. Good internal consistency and concurrent validity with the Clinician-assessed PTSD Scale.
Change in Beck Anxiety Inventory | Baseline (pre-treatment), Every session (weekly) if primary /target problem up to 16 weeks
  21-item self-report instrument for measuring the severity of anxiety symptoms. Good internal consistency (α = .92) and high test-retest reliability (r = .75.).

SECONDARY OUTCOMES:
Change in Inventory of Psycho social Functioning-Brief Version | Completed at baseline, One Month, and post-treatment (week 16)
  14 items, yields a grand mean and 7 subscale means for functioning in romance, family, friendships, parenting, education, work, and self-care activities (non-applicable categories can be skipped; total score reflects mean of applicable items). Excellent reliability and internal consistency ( α = 0.93); correlates with other measures of quality of life.
Evidence-Based Practice Attitudes Scale-50 (EBPAS) | Completed at therapist baseline (prior to providing treatment in the study)
  This measure looks at Evidence-based practice attitudes and motivation among clinicians, 1 (worse)-5 (best) total score range
Perceived Characteristics of Interventions (PCIS) | Completed at therapist baseline (prior to providing treatment in the study)
  Innovation characteristics hypothesized to influence adoption and sustainability
Implementation Climate Assessment (ICA) | Completed at therapist baseline (prior to providing treatment in the study)
  Brief validated measure of implementation climate ( manager support for EBPs, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon W Stirman, PhD, Principal Investigator — NCPTSD/Stanford University
Locations (4):
- United States (4):
  - VA Palo Alto Health Care System, Palo Alto, California
  - NCPTSD - VA Boston HCS, Boston, Massachusetts
  - Massachusetts General Hospital, Chelsea, Massachusetts
  - Aaron T. Beck Psychopathology Research Center, Philadelphia, Pennsylvania

REFERENCES:
- [Background] McHugh RK, Barlow DH. The dissemination and implementation of evidence-based psychological treatments. A review of current efforts. Am Psychol. 2010 Feb-Mar;65(2):73-84. doi: 10.1037/a0018121. PMID 20141263
- [Background] Schoenwald SK. It's a Bird, It's A Plane, It's ... Fidelity Measurement In the Real World. Clin Psychol (New York). 2011 Jun;18(2):142-147. doi: 10.1111/j.1468-2850.2011.01245.x. PMID 21691439
- [Background] Schoenwald SK, Garland AF, Chapman JE, Frazier SL, Sheidow AJ, Southam-Gerow MA. Toward the effective and efficient measurement of implementation fidelity. Adm Policy Ment Health. 2011 Jan;38(1):32-43. doi: 10.1007/s10488-010-0321-0. PMID 20957425
- [Background] Ruzek JI, Rosen RC. Disseminating evidence-based treatments for PTSD in organizational settings: A high priority focus area. Behav Res Ther. 2009 Nov;47(11):980-9. doi: 10.1016/j.brat.2009.07.008. Epub 2009 Jul 26. PMID 19632668
- [Background] Carroll KM, Martino S, Rounsaville BJ. No train, no gain? Clinical Psychology: Science and Practice. 2010;17(1):36-40.
- [Background] Decker SE, Jameson MT, Naugle AE. Therapist training in empirically supported treatments: a review of evaluation methods for short- and long-term outcomes. Adm Policy Ment Health. 2011 Jul;38(4):254-86. doi: 10.1007/s10488-011-0360-1. PMID 21656256
- [Background] Resick PA, Galovski TE, Uhlmansiek MO, Scher CD, Clum GA, Young-Xu Y. A randomized clinical trial to dismantle components of cognitive processing therapy for posttraumatic stress disorder in female victims of interpersonal violence. J Consult Clin Psychol. 2008 Apr;76(2):243-258. doi: 10.1037/0022-006X.76.2.243. PMID 18377121
- [Background] Resick PA, Monson CM, Chard KM. Cognitive processing therapy veteran/military version: Therapist and patient materials manual. . Washington, DC: Department of Veterans' Affairs; 2008.
- [Background] Beck AT. The current state of cognitive therapy: a 40-year retrospective. Arch Gen Psychiatry. 2005 Sep;62(9):953-9. doi: 10.1001/archpsyc.62.9.953. PMID 16143727
- [Background] Clark DM. Implementing NICE guidelines for the psychological treatment of depression and anxiety disorders: the IAPT experience. Int Rev Psychiatry. 2011 Aug;23(4):318-27. doi: 10.3109/09540261.2011.606803. PMID 22026487
- [Background] Karlin BE, Cross G. From the laboratory to the therapy room: National dissemination and implementation of evidence-based psychotherapies in the U.S. Department of Veterans Affairs Health Care System. Am Psychol. 2014 Jan;69(1):19-33. doi: 10.1037/a0033888. Epub 2013 Sep 2. PMID 24001035
- [Background] Karlin BE, Ruzek JI, Chard KM, Eftekhari A, Monson CM, Hembree EA, Resick PA, Foa EB. Dissemination of evidence-based psychological treatments for posttraumatic stress disorder in the Veterans Health Administration. J Trauma Stress. 2010 Dec;23(6):663-73. doi: 10.1002/jts.20588. Epub 2010 Nov 15. PMID 21171126
- [Background] Foa EB, Keane TM, Friedman MJ, Cohen JA. Effective treatments for PTSD: Practice guidelines from the International Society for Traumatic Stress Studies (2nd ed.). New York, NY US: Guilford Press; 2009.
- [Background] Stirman SW, Buchhofer R, McLaulin JB, Evans AC, Beck AT. Public-academic partnerships: the Beck Initiative: a partnership to implement cognitive therapy in a community behavioral health system. Psychiatr Serv. 2009 Oct;60(10):1302-4. doi: 10.1176/ps.2009.60.10.1302. PMID 19797367
- [Background] Mendel P, Meredith LS, Schoenbaum M, Sherbourne CD, Wells KB. Interventions in organizational and community context: a framework for building evidence on dissemination and implementation in health services research. Adm Policy Ment Health. 2008 Mar;35(1-2):21-37. doi: 10.1007/s10488-007-0144-9. Epub 2007 Nov 8. PMID 17990095
- [Background] Chambers DA, Glasgow RE, Stange KC. The dynamic sustainability framework: addressing the paradox of sustainment amid ongoing change. Implement Sci. 2013 Oct 2;8:117. doi: 10.1186/1748-5908-8-117. PMID 24088228
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Beck AT, Steer RA. Manual for the Beck anxiety inventory. 1990.
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Derived] Calloway A, Creed TA, Gumport NB, Gutner C, Marques L, Hernandez S, Song J, Johnson C, Youn SJ, Elhusseini S, Deguzman-Lucero RM, Laskot T, La Bash H, Silvan YA, Cassotte C, Park AL, Dean K, Bartuska AD, Jo B, Barnett P, Kuhn E, DeRubeis R, Vogt D, Stirman SW. A comparison of scalable routine clinical materials and observer ratings to assess CBT fidelity. Behav Res Ther. 2025 Jan;184:104655. doi: 10.1016/j.brat.2024.104655. Epub 2024 Nov 26. PMID 39612724
- [Derived] Wiltsey Stirman S, Marques L, Creed TA, Gutner CA, DeRubeis R, Barnett PG, Kuhn E, Suvak M, Owen J, Vogt D, Jo B, Schoenwald S, Johnson C, Mallard K, Beristianos M, La Bash H. Leveraging routine clinical materials and mobile technology to assess CBT fidelity: the Innovative Methods to Assess Psychotherapy Practices (imAPP) study. Implement Sci. 2018 May 22;13(1):69. doi: 10.1186/s13012-018-0756-3. PMID 29789017